CLINICAL TRIAL: NCT02148705
Title: A Multicenter, Multinational, Randomized, Controlled, Assessor Blinded Study, Performed in Subjects With Thermal Burns, to Evaluate the Efficacy and Safety of NexoBrid Compared to Gel Vehicle and Compared to Standard of Care
Brief Title: A Study to Evaluate the Efficacy and Safety of NexoBrid in Subjects With Thermal Burns
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MW 2010-03-02
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-06

CONDITIONS: Thermal Burns
Keywords: fire/flame; scalds; contact
MeSH Terms: interventions — Standard of Care; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NexoBrid Gel (Experimental): NexoBrid Gel is applied to the burn wound at a dose of 2 g NexoBrid sterile powder mixed with 20g sterile Gel Vehicle per 1% of TBSA (~ surface of an adult palm) for four hours.
  Interventions: Drug: NexoBrid
- Gel Vehicle (Placebo Comparator): Gel Vehicle is applied to the burn wound at a dose of 20 g sterile Gel per 1% of TBSA (~ surface of an adult palm) for four hours.
  Interventions: Drug: Gel Vehicle
- Standard of Care (SOC) (Active Comparator): Subjects in the SOC group may be treated with a combination of surgical and non-surgical eschar removal procedures, according to the investigator's judgment.
  Interventions: Procedure: Standard of Care (SOC)

INTERVENTIONS:
Drug: NexoBrid
  Arms: NexoBrid Gel
Procedure: Standard of Care (SOC)
  Arms: Standard of Care (SOC)
Drug: Gel Vehicle
  Arms: Gel Vehicle

SUMMARY:
This study will be a three-arms study intending to demonstrate superiority of NexoBrid treatment over the Gel Vehicle placebo control treatment and over SOC in thermal burn subjects.

The study objectives are:

1. To demonstrate the efficacy of enzymatic eschar removal with NexoBrid by providing complete eschar removal as compared with Gel vehicle,
2. To demonstrate the efficacy of enzymatic eschar removal with NexoBrid by providing earlier complete eschar removal, reduction in patients' surgical burden and its related blood loss as compared to SOC,
3. To assess the safety of NexoBrid compared to SOC, including demonstration that treatment with NexoBrid does not cause an unacceptable level of harm on wound closure outcome and long term outcomes of cosmesis and function.

DETAILED DESCRIPTION:
This is a multi-center, multi-national, randomized, controlled, assessor blinded, three-arm study aiming to demonstrate superiority of NexoBrid treatment over Gel Vehicle control and over SOC treatment in thermal burn subjects with burns. Following the enrollment of a patient to the study and prior to randomization Physicians will define one or more Target Wounds (TWs) per subject according to TWs definition. All subjects' deep (DPT and FT) burns that comply with the specified entrance criteria are intended to receive study treatment per the randomized study arm.

The randomization procedure will be initiated only after all Target wounds of a subject have been defined. Patients will be assigned to the treatment arm in a 3:3:1 ratio (NexoBrid: SOC : Gel Vehicle).

Patients will be treated in the same way in all study arms (NexoBrid, SOC or Gel vehicle) except for the eschar removal stage which will be performed as per the randomization study arm.

Prior to initiation of eschar removal treatment, subjects will be medicated with appropriate analgesia and undergo wound cleansing and dressing of all wounds with antibacterial solutions . Following wound cleansing and antibacterial treatments, subjects will undergo the eschar removal process as per treatment assignment (NexoBrid, SOC or Gel Vehicle, following randomization).

Subsequent to complete eschar removal, all wounds will be assessed and treated in the same manner, in accordance with post-eschar removal wound care strategy. Post eschar removal, subjects will undergo daily vital signs and pain assessments, until hospital discharge (HD) and weekly assessments of wound progress, until wound closure. Following wound closure confirmation visit, subjects will be followed up at 1, 3, 6, 12, 18 and 24 months post wound closure for long term outcomes evaluation.

ELIGIBILITY:
Inclusion Criteria- Patient level

1. Males and females; ≥ 18
2. Thermal burns caused by fire/flame, scalds or contact,
3. Patient total burns area ≥ 3% DPT and / or FT,
4. Patient total burns area should be ≤ 30% TBSA; SPT, DPT and/or FT in depth,
5. Informed consent can be obtained within 84 hours of the burn injury,
6. Patients who are willing and able to sign a written consent form.

Inclusion Criteria - Wound level

1. At least one wound (a continuous burn area) that is ≥0.5% TBSA (DPT and/or FT) (this minimal wound size should not including face, perineal or genital area.

   All planned target wounds (TWs) should meet the following criteria:
2. SPT area that cannot be demarcated from DPT and FT areas should be less than 50% of the % TBSA of the TW.
3. Wound's blisters can be removed/ unroofed, as judged by the investigator.

Exclusion Criteria- Patient level

1. Patients who are unable to follow study procedures and follow up period.
2. Modified Baux index ≥ 80,
3. Patients with burned charred fingers, 3rd degree in depth and possibly devoid of circulation,
4. Patients with abraded wound/s that cannot be treated by an enzymatic debrider application (NexoBrid) will be excluded from the study,
5. Patients with electrical or chemical burns,
6. Patients with circumferential (≥ 80% of the limb circumference) DPT and/or FT burns defined as Extremities at Risk (EAR) 2 as described in the protocol.
7. The following pre-enrollment dressings: a. Flammacerium, b. Silver Nitrate (AgNO3),
8. Patients with pre-enrolment wounds which are covered by eschar heavily saturated with iodine or by SSD pseudoeschar (e.g. pseudoeschar as a result of > 12 hours SSD treatment),
9. Patients with pre-enrollment escharotomy.
10. Patients with diagnosed infections as described in Section 11.9 of study protocol,
11. Diagnosis of smoke inhalation injury.
12. Pregnant women (positive pregnancy test) or nursing mothers.
13. Poorly controlled diabetes mellitus (HbA1c>11%) in patients with known diabetes as captured in the medical history.
14. BMI greater than 39.0 kg/m2 in patients with burn area up to 15% TBSA or BMI greater than 34.0 kg/m2 in patients with burn area more than 15% TBSA.
15. ASA greater than 2 (Appendix 13- ASA classification system)
16. Cardio-pulmonary disease (MI within 6 months prior to injury, severe pulmonary hypertension, severe COPD or pre-existing oxygen-dependent pulmonary diseases, severe broncho-pneumonia within 1 month prior to injury , steroid dependent asthma or uncontrolled asthma).
17. Pre-existing diseases which interfere with circulation (severe peripheral vascular disease, edema, lymphedema, regional lymph nodes, significant varicose veins),
18. Any conditions that would preclude safe participation in the study or adding further risk to the basic acute burn trauma (such as severe immuno-compromising diseases, life threatening trauma, severe pre-existing coagulation disorder,severe cardiovascular disorder,significant pulmonary disorder, significant liver disorder including post alcoholic abuse impaired function or neoplastic disease, blast injury)
19. Chronic systemic steroid intake,
20. History of allergy and/or known sensitivity to pineapples, papaya, Bromelain or papain,
21. Current (within 12 months prior to screening) suicide attempt,
22. Mentally incapacitated adults who are incapable of giving legal consent
23. Enrollment in any investigational drug trial within 4 weeks prior to screening,
24. Current (within 12 months prior to screening) alcohol or drug abuse (see definition in section 1.1)
25. Prisoners and incarcerated,
26. Patients who might depend on the clinical study site or investigator.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (18):
  - University of South Alabama Department of Surgery, Mobile, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - University of Colorado at Denver, Teaching, Aurora, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida- Dept. of Surgery, Gainesville, Florida
  - Joseph M. Still Research Foundation, Inc., Augusta, Georgia
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Burnett Burn Center at The University of Kansas Hospital, Kansas City, Kansas
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - The General Hospital Corporation d/b/a Massachusetts General Hospital, Boston, Massachusetts
  - New-York Presbyterian Hospital, New York, New York
  - Emergency Medicine Stony Brook University Hospital, Stony Brook, New York
  - Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania
  - Regional Medical Center ,Regional One Health, Memphis, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - HarborView Medical Center, Seattle, Washington
  - Columbia St. Mary's, Inc., Milwaukee, Wisconsin
- University Hospital, Department of Plastic Surgery, Ghent, Belgium
- Klinika popálenin a rekonstrukční chirurgie, Fakultní nemocnice Brno, Brno, Czechia
- Khechinashvili University Hospital - Thermal Injuries, Tbilisi, Georgia
- Germany (2):
  - Unfallkrankenhaus Berlin Zentrum für Schwerbrandverletzte mit Plastischer Chirurgie, Berlin
  - BG Universitätsklinikum Bergmannsheil GmbH, Bochum
- Rambam Medical Center, Haifa, Israel
- Italy (2):
  - Hospital A. Cardarelli of Napoli, Napoli
  - Ospedale di Cisanello, Pisa
- Romania (3):
  - Spitalul Clinic de Urgenta de Chirurgie Plastica, Reparatorie si Arsuri, Bucharest
  - Spitalul Clinic de Urgenta "Sf. Ioan", Bucharest
  - Spitalul Clinic de Urgenta "Bagdasar-Arseni", Bucharest

REFERENCES:
- [Derived] Shoham Y, Rosenberg L, Hickerson W, Goverman J, Iyer N, Barrera-Oro J, Lipovy B, Monstrey S, Blome-Eberwein S, Wibbenmeyer LA, Scharpenberg M, Singer AJ. Early Enzymatic Burn Debridement: Results of the DETECT Multicenter Randomized Controlled Trial. J Burn Care Res. 2024 Mar 4;45(2):297-307. doi: 10.1093/jbcr/irad142. PMID 37715999

RESULTS

PARTICIPANT FLOW:
Groups:
- NexoBrid Gel: NexoBrid Gel is applied to the burn wound at a dose of 2 g NexoBrid sterile powder mixed with 20g sterile Gel Vehicle per 1% of TBSA (~ surface of an adult palm) for four hours.
  NexoBrid
- Gel Vehicle: Gel Vehicle is applied to the burn wound at a dose of 20 g sterile Gel per 1% of TBSA (~ surface of an adult palm) for four hours.
  Gel Vehicle
- Standard of Care (SOC): Subjects in the SOC group may be treated with a combination of surgical and non-surgical eschar removal procedures, according to the investigator's judgment.
  Standard of Care (SOC)
Period: Overall Study
Arm/Group | NexoBrid Gel | Gel Vehicle | Standard of Care (SOC)
Started | 75 | 25 | 75
Treated | 77 (Two patients randomized to SOC were treated with NexoBrid and are included in the safety (treated) population) | 24 | 68
Completed Acute Phase | 67 | 23 | 63
Completed 12M FU Period | 57 | 20 | 58
Completed | 57 | 20 | 58
Not Completed | 18 | 5 | 17
Not completed — Death | 2 | 0 | 0
Not completed — Lost to Follow-up | 13 | 4 | 10
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — Not Treated | 0 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Overall 175 randomized patients are the baseline participants (Full Analysis Set, FAS). Out of the 175, 169 were treated (safety population): 77 In NexoBrid Gel arm, 24 In Gel Vehicle arm (Placebo) and 68 in the SOC arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | NexoBrid Gel | Gel Vehicle | Standard of Care (SOC) | Total
Number analyzed (Participants) | 75 | 25 | 75 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 21 | 70 | 159
  >=65 years | 7 | 4 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.28 (15.03) | 40.68 (17.30) | 40.91 (15.16) | 40.95 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 16 | 52
  Male | 49 | 15 | 59 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 8 | 8 | 30
  Not Hispanic or Latino | 61 | 17 | 67 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 3 | 13 | 24
  White | 61 | 21 | 59 | 141
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Number of Participants With Complete Eschar Removal.
Description: Comparison of NexoBrid over Gel Vehicle for eschar removal as measured by Number of Participants with complete eschar removal at the end of the topical agent soaking period by a blinded assessor.
Time Frame: post application (post 2 h soaking)
Population: Standard of Care (SOC) is not included as it was pre-specified in the statistical analysis plan that for the primary endpoint, NexoBrid Gel will be compared only to the Gel Vehicle
Measure: Count of Participants; unit: Participants
Arm/Group | NexoBrid Gel | Gel Vehicle
Number analyzed (Participants) | 75 | 25
Participants | 70 | 1
Statistical Analysis 1: Comparison: NexoBrid Gel vs Gel Vehicle; Test type: Superiority; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 288.281, 95% CI 2-sided [35.549 to 13984.356]

2. Secondary Outcome: Secondary Endpoint: Number of Participants With Surgical Excision Performed or Eschar Removal for NexoBrid vs SOC (FAS)
Description: Comparison of NexoBrid over SOC in number of Participants with surgical need for excisional eschar removal as measured by an analysis of incidence of surgical eschar removal (tangential/ minor/ avulsion/ Versajet and/or dermabrasion excision).
Time Frame: Post application (post 2 h soaking) for NexoBrid arm and immediately post surgical excision for SOC arm.
Population: Gel arm is not involved in comparison as defined in the statistical analysis plan. Only NexoBrid and SOC
Measure: Count of Participants; unit: Participants
Arm/Group | NexoBrid Gel | Standard of Care (SOC)
Number analyzed (Participants) | 75 | 75
Participants | 3 | 54
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care (SOC); Test type: Superiority; p < 0.0001, Chi-squared; Odds Ratio (OR) = 0.011, 95% CI 2-sided [0.003 to 0.044]

3. Secondary Outcome: Secondary Endpoint: Comparison of Time (Days) to Complete Eschar Removal
Description: Comparison of NexoBrid over SOC with regard to the time (in days) when complete eschar removal has been achieved. Results of the Generalized Wilcoxon-Gehan Test Adjusted for Overall TW Depths, TBSA Group, Center Group, and Number of TWs (FAS)
Time Frame: From randomization until complete eschar removal. For NexoBrid, assessed post application (post 2 h soaking) and for SOC assessed immediately post last dressing change for non-surgical SOC arm and immediately post excision for surgical SOC arm.
Population: Gel arm is not involved in comparison as defined in the statistical analysis plan. Only NexoBrid and SOC
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NexoBrid Gel | Standard of Care (SOC)
Number analyzed (Participants) | 75 | 75
Days | 1.02 [0.98 to 1.07] | 3.87 [1.98 to 5.98]
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care (SOC); Test type: Superiority; p < 0.0001, Generalized Wilcoxon-Gehan Test; Analysis is adjusted for Overall TW Depths, TBSA Group, Center Group, and Number of TWs; Test Statistics = 23.1429

4. Secondary Outcome: Secondary Endpoint: Patient-Level Comparison of Actual Blood Loss (Volume in mL) Related to Eschar Removal for NexoBrid vs SOC (FAS)
Description: Comparison of NexoBrid over SOC with regard to the blood loss (volume in mL) occurred during the eschar removal procedures.
Time Frame: For NexoBrid arm, blood loss during NexoBrid application until post soaking. For SOC arm, blood loss during SOC procedures, through last dressing change for non-surgical SOC arm and through excision surgery for surgical SOC arm.
Population: Gel arm is not involved in comparison as defined in the statistical analysis plan. Only NexoBrid and SOC were compared
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NexoBrid Gel | Standard of Care (SOC)
Number analyzed (Participants) | 75 | 75
mL | 14.17 (512.40) | 814.51 (1020.32)
Statistical Analysis 1: Comparison: NexoBrid Gel vs Standard of Care (SOC); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon tests pooled using Rubin´s rule; estimate = 6505.80, 95% CI 2-sided [5974.41 to 7037.19], Standard Error of Mean 269.88

ADVERSE EVENTS:
Time Frame: Time of informed consented until subject's study completion (12 months post wound closure) or earlier if early termination from study.
Description: An adverse event is an undesirable or unintentional event that occurs during use of the study Drug, whether or not considered related to the Drug; this includes clinically significant changes in laboratory values and therapeutic failures. Regardless of the severity or relationship to the investigational Drug, all adverse events occurring during the study period should be recorded in a subject's CRFs.
Arm/Group | NexoBrid Gel | Gel Vehicle | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 2/77 | 0/24 | 0/68
Serious Adverse Events (participants affected / at risk) | 9/77 | 3/24 | 9/68
Other Adverse Events (participants affected / at risk) | 49/77 | 16/24 | 39/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NexoBrid Gel (N=77) | Gel Vehicle (N=24) | Standard of Care (SOC) (N=68)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Congenital Tricuspid Valve Incompetence (Congenital, familial and genetic disorders) | 1 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 1 | 0 | 0
Persistent Fetal Circulation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 1 | 0 | 0
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma of the Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral Ventricle Dilatation (Nervous system disorders) | 1 | 0 | 0
Failure to Thrive (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Neonatal Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Transient Tachypnoea of the Newborn (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eventration Repair (Surgical and medical procedures) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Acute Coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Bifascicular Block (Cardiac disorders) | 0 | 0 | 1
Appendicitis Noninfective (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Infusion Site Thrombosis (General disorders) | 0 | 1 | 0
Wound Infection Bacterial (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft Loss (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Internal Fixation of Fracture (Surgical and medical procedures) | 1 | 0 | 0
Therapeutic Procedure (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 1
Phlebitis Superficial (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NexoBrid Gel (N=77) | Gel Vehicle (N=24) | Standard of Care (SOC) (N=68)
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 2
Vomiting (Gastrointestinal disorders) | 5 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 2 | 6
Pyrexia (General disorders) | 4 | 2 | 5
Pain (General disorders) | 4 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 0 | 0
Wound Infection Bacterial (Infections and infestations) | 4 | 0 | 4
Sepsis (Infections and infestations) | 3 | 0 | 0
Sinusitus (Infections and infestations) | 1 | 1 | 3
Graft Loss (Injury, poisoning and procedural complications) | 3 | 1 | 3
Wound Complications (Injury, poisoning and procedural complications) | 3 | 0 | 2
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 6 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (8):
  • Study Protocol: Protocol version 11 (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/Prot_000.pdf
  • Study Protocol: Protocol Version 9 (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/Prot_001.pdf
  • Study Protocol: Protocol Version 8 (2015-02-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/Prot_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Protocol V11 V3amendment 02 (2020-08-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/SAP_003.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Protocol V11 V3amendment 01 (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/SAP_004.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Protocol V11 V3 (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/SAP_005.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Protocol V11 V2amendment 01 (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/SAP_006.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Protocol V11 V2 (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT02148705/SAP_007.pdf